CLINICAL TRIAL: NCT01655849
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate The Efficacy and Safety of Z160 in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Brief Title: Phase 2 Efficacy Trial of Z160 in Lumbosacral Radiculopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z160-LSR-201
Record Dates: First submitted 2012-07-26; First posted 2012-08-02 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Lumbosacral Radiculopathy
MeSH Terms: interventions — Z160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z160 (Experimental): 375mg BID
  Interventions: Drug: z160
- placebo (Placebo Comparator): matching placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: z160
  Arms: Z160
Drug: Placebo
  Arms: placebo

SUMMARY:
This study will compare Z160 and placebo in patients with Lumbosacral Radiculopathy for safety and efficacy for a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have a diagnosis of pain due to LSR, with all of the following characteristics:

   * The subject perceives pain in one or both lower limbs at sites that are consistent with the area innervated by the L4, L5, or S1 nerve roots, with or without other sensory symptoms in the affected areas (typically, the pain may be perceived in the buttock, thigh, calf, leg, foot, or toes).
   * The history of the pain suggests that the cause of the LSR is due to injury of the lumbosacral nerve root(s) by degenerative disease of the vertebrae in the lumbosacral spine or associated soft tissues (including the intervertebral discs).
   * The duration of pain since onset is ≥ 12 weeks.
   * Based on clinical history, the intensity of pain has been stable during the 2-week period before screening.
2. In the investigator's opinion, the subject's diagnosis of LSR is supported by all of the following at screening:

   * Based on the StEP instrument:

     * Neurological examination of lower limbs shows impaired muscle power, sensory function, or deep tendon reflexes in the territory of the affected nerve roots.
     * Pain/sensory disturbance in dermatomal/myotomal distribution is precipitated or exacerbated by straight leg raising (the straight-leg-raising test should be performed as specified in StEP).
     * The total StEP score is ≥ 4 (indicative of LSR as the cause of the pain)

4. At screening, the subject has an average daily pain score for neuropathic pain due to LSR of ≥ 3 and ≤ 8 on the PI-NRS.

5. If female, the subject must be postmenopausal (defined as no menstruation for at least 12 months), surgically sterilized for ≥3 months before the screening visit, or agree to use 2 reliable methods of contraception (oral, implantable, transdermal, or injectable contraceptives in conjunction with an intrauterine device or a barrier method) during the 6-week treatment period, during the 6 week posttreatment follow-up period, and for an additional 8 weeks after the last study visit (Week 12, Visit 9) to avoid pregnancy if of childbearing potential (defined as biologically capable of becoming pregnant). If male, the subject must agree to use condoms during the 6-week treatment period with the study drug, during the 6-week posttreatment follow up period, and for an additional 8 weeks after the last study visit (Week 12, Visit 9).

Exclusion Criteria:

1. The subject has:

   * Neuropathic pain due to causes other than that specified in the inclusion criteria (e.g., postherpetic neuralgia; painful diabetic neuropathy; mononeuritis multiplex; central poststroke pain; failed back surgery in relation to the presenting episode of radiculopathy; spinal abscess, infection, hematoma, or malignancy; phantom limb pain; peripheral neuropathy due to alcoholism, malignancy, human immunodeficiency virus [HIV], syphilis; drug abuse; vitamin B12 deficiency; hypothyroidism; liver disease; toxic exposure).
   * Pain that is associated with a substantial somatic pain component (e.g., non-neuropathic/musculoskeletal pain in lower limbs or other parts of the body apart from the back) or more than one cause or potential cause for pain symptoms.
   * Any painful concurrent rheumatic disease such as, but not limited to, fibromyalgia, rheumatoid arthritis, or significant osteoarthritis.

   Any question regarding the acceptability of the etiology of the neuropathic pain should be discussed with the Zalicus medical monitor.
2. In the investigator's opinion, the subject is unable to reliably delineate or assess his or her own pain by anatomical location/distribution (e.g., the subject cannot reliably tell the difference between his or her back pain and lower limb pain and cannot rate the intensity of each separately).
3. The subject has pain in the lower limbs solely upon walking and not at rest.
4. The subject has undergone surgery for LSR within the last 6 months or has received treatment with epidural injections, nerve blocks, or acupuncture for LSR within 4 weeks before screening.
5. The subject has:

   * A history of seizure, excluding pediatric febrile seizures, or currently has seizures
   * A history of or a current diagnosis of schizophrenia or bipolar disorder
   * Had a stroke or TIA ≤ 6 months before the screening visit
   * Has an episode of major depression or generalized anxiety disorder ≤ 6 months before the screening visit.
6. The subject has a history of or currently has any of the following conditions that, in the investigator's opinion, may interfere with the study procedures or compromise the subject's safety:

   * Cardiovascular disease
   * Gastrointestinal disease
   * Hepatic disease
   * Respiratory disease
   * Renal disease
   * Any condition that is known to interfere with the absorption, distribution, metabolism, or excretion of drugs
7. The subject has a history of or currently has:

   * Any clinically significant vital sign, ECG, or laboratory abnormalities.
   * QTcF >450 msec (males) or >470 msec (females)
8. The subject had a malignancy.
9. The subject has had a positive test for HIV antibody or a history of HIV.
10. The subject has had a positive test for hepatitis B surface antigen or hepatitis C antibody.
11. The subject has a history of AST, ALT or bilirubine >2 times the upper limit of normal.
12. The subject has a history of hypersensitivity to calcium channel blockers.
13. The subject has a history of multiple drug allergies (≥ 2 kinds) that, in the investigator's opinion, may place him or her at greater risk during participation in the study.
14. The subject has participated in a previous clinical study of Z160 or has received another investigational drug ≤ 30 days before the screening visit.
15. The subject has taken a prohibited medication ≤ 30 days before the screening visit.
16. The subject has a history of alcohol or narcotic substance abuse, as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), ≤ 1 year before the screening visit.
17. The subject has a positive urine drug test at screening.
18. The subject is female and is pregnant or breastfeeding at the time of the screening visit or plans to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in weekly average of daily pain scores (PI-NRS) | Baseline to week 6

SECONDARY OUTCOMES:
Change in weekly average of daily pain scores (PI-NRS) | Baseline to weeks 1,2,3,4,5, 6
Galer Neuropathic Pain Scale (NPS) | Baseline to weeks 1,2,4,6
Patient Global Impression of Change (PGIC) | Baseline to week 6
Modified Roland-Morris Disability Scale (RMDQ) | Baseline to weeks 1,2,4,6
Rescue medication use | Weeks 1,2,3,4,5,6
Profile of Mood States (POMS) | Baseline to weeks 1,2,4,6
Daily Sleep Interference Scale | Baseline to weeks 1,2,3,4,5,6
Short Form 36 (SF-36) | Baseline to week 6
Safety and tolerability | Baseline, weeks 1,2,3,4,5,6,7,12
  Adverse events, ECG, labs
Relationship of plasma concentrations | Baseline to weeks 1,2,3,4,5,6
Time to a 30% reduction in average daily pain score | Baseline to weeks 1,2,3,4,5,6
Time to a 50% reduction in average daily pain score | Baseline to weeks 1,2,3,4,5,6
Subjects who have greater than or equal to a 30% reduction in average daily pain score | Baseline to weeks 1,2,3,4,5,6
Subjects who have greater than or equal to a 50% reduction in average daily pain score | Baseline to weeks 1,2,3,4,5,6

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lee, PhD, Study Director — Zalicus Inc
Locations (22):
- United States (22):
  - Investigative Site, Huntsville, Alabama
  - Investigative Site, Peoria, Arizona
  - Investigative Site, Anaheim, California
  - Investigative Site, Fresno, California
  - Investigative Site, Orange, California
  - Investigative Site, Sacramento, California
  - Investigative Site, Clearwater, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Pinellas Park, Florida
  - Investigative Site, Plantation, Florida
  - Investigative Site, Royal Palm Beach, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Hazelwood, Missouri
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, Medford, Oregon
  - Investigative Site, Duncansville, Pennsylvania
  - Investigative Site, Dallas, Texas
  - Investigative Site, Sandy City, Utah
  - Investigative Site, Bellevue, Washington